CLINICAL TRIAL: NCT01443806
Title: Characterisation of the Human Carboxylesterase 1 (CES1) Mutation(s) Which May be Responsible for Markedly Reduced Conversion of Oseltamivir Phosphate to Oseltamivir Carboxylate
Brief Title: Characterisation of the Human Carboxylesterase 1 (CES1) Mutations in Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: South East Asia Infectious Disease Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SEA 026
Record Dates: First submitted 2011-07-12; First posted 2011-09-30 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Disease
Keywords: oseltamivir metabolism; Carboxylesterase 1
MeSH Terms: conditions — Metabolic Diseases | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oseltamivir, genetic testing (Experimental)
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — 75 mg, one time
  Other Names: Tamiflu

SUMMARY:
The aim of this study is to evaluate the conversion of OP to OC in individual X and the family member of individual X. The investigators hypothesize that one or more of the single nucleoprotein polymorphisms (SNPs) of the CES1 gene represent a clinically important functional polymorphism.

DETAILED DESCRIPTION:
Oseltamivir is beneficial in the treatment of mild influenza. When given by mouth, oseltamivir phosphate (OP), the parent drug, is rapidly absorbed and rapidly converted to oseltamivir carboxylate (OC) by carboxylesterase enzymes (CES1) in the gut, plasma and liver. The mean time to maximum concentration of OP is 2 hours and OC is about 4. Plasma protein binding is ~42% for OP and <3% for OC. The latter has a volume of distribution at steady state after an IV dose of 23 to 26 L which is similar to extracellular water, consistent with its polar nature and low protein binding. OC and OP are renally excreted via glomerular filtration and active secretion via the organic anion transporter in the proximal renal tubules. In healthy subjects, oseltamivir carboxylate has a half life of 6-11 hours, achieves steady-state within 3 days (bd dosing) and has a higher AUC on Day 7 compared to Day 1.

Oseltamivir was associated with bizarre behaviour and acute confusion. Since these reports, similar events have also been associated with inhaled zanamivir, suggesting that the influenza rather than the drugs were responsible.

Because OP is more lipophilic than OC, it should cross the blood brain barrier more easily than OC. However, plasma to CSF ratios in 4 healthy volunteers were low for both substances, just over two and just under 3.5% for OP and OC, respectively. The low OP ratio is probably due to the actively export of OC from the brain by P-glycoprotein pump. In vitro and mice studies demonstrate that OP but not OC is a substrate for the glycoprotein P (P-gp) transporter and that the brain distribution of OC is affected by P-gp activity. PK simulations predict levels of OP that would be within the range of exposures observed in clinical studies without neuropsychiatric adverse effects.

One individual subject (individual X) from SEA004 "Long Term Influenza Prophylaxis with Inhaled Zanamivir or Oral Oseltamivir" had carboxylesterase 1 (CES1) gene mutation which may affect oseltamivir phosphate conversion. This means that the conversion of OP to OC in this subject can be substantially lower than the normal population.

This is a very important finding relevant both to antiviral efficacy and also potentially to toxicity because OP has no antiviral activity and may play a role in toxicity as a potentially neuroexcitatory compound. On the basis of in vitro data, the risk of cardiac toxicity should be not existent at therapeutic doses. OP had a variable effect on the hERG (human ether a go go K+ channel in cardiac muscle) but only at concentrations far in excess of those achieved with therapeutic doses; OC has no proarrhythmic effect.

Given that OP penetrates the blood brain barrier and is pumped out by P-glycoprotein, high plasma concentrations of OP could result in increased CNS concentrations in individuals with either reduced carboxylesterase activity, such as infants and the volunteer in this study and/or reduced P-glycoprotein activity.

Human carboxylesterase 1 (CES1) polymorphisms CES1 is a member of a multigene family of serine esterases that is involved in drug metabolism and activation as well as in other biological processes. The study from Shi et al reported the correlation between oseltamivir hydrolysis from OP to OC and the concentration of CES1.

The gene encoding CES1 is on the long arm of chromosome 16 (16q13-22.1), and consists of 14 exons spanning 30kb. Several studies have identified the CES1 gene polymorphisms in the promoter and coding region and have tried to relate these polymorphisms with variation in the hydrolysis activity of this protein. A study from Zhu HJ et al presented potentially 2 functional polymorphisms locating in exon 4 (Gly143Glu) and 6 (Asp260fs) that can impair the CES1 hydrolytic activity to methylphenidate in vitro. However, some CES1 variants (V21I, and R182H) have a higher rate of oseltamivir metabolism compared to wild-type.

All subjects from these reports were recruited from Japanese and European populations. Therefore, it would be important to investigate the CES1 gene in the Thai population.

Oseltamivir efficacy may well be compromised in individuals who do not convert OP to OC but there are no data on the prevalence of this mutation/polymorphism and, therefore, the number of individuals who may not benefit form oseltamivir is unknown.

It will be important to study further the carboxylesterase gene in order to characterise its inheritance in the family of individual X and then to conduct prevalent studies in e.g. stored serum banks and as part of PK studies of oseltamivir in patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy family member of individual X and individual X
* Aged between 18 and 70, inclusive.

Exclusion Criteria:

* known allergy to oseltamivir
* any underlying illness that is considered a risk to the health of the individual
* pregnant
* breast feeding
* creatinine clearance < 30 mL/min calculated by the Cockcroft Gault formula: CrCl (ml/min) = (140-age) x Wt in kg / creatinine mg/dL x 72, for females, the result is multiplied by 0.85.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tmax | 2 and 4 hours
  Conversion of Oseltamivir at 2 and 4 hours post dose

SECONDARY OUTCOMES:
Conversion of oseltamivir phosphate to oseltamivir carboxylate | one year (anticipate)
  Document the sequence of all 14 exons of CES1 from individual X and the family members of individual X.

CONTACTS AND LOCATIONS:
Overall Officials: Sasithon Pukrittayakamee, MD., Principal Investigator — Mahidol University
Locations (1):
- The Faculty of Tropical medicine,Mahidol University, Bangkok, Thailand